CLINICAL TRIAL: NCT03153579
Title: LSD Treatment in Persons Suffering From Anxiety Symptoms in Severe Somatic Diseases or in Psychiatric Anxiety Disorders: a Randomized, Double-blind, Placebo-controlled Phase II Study
Brief Title: LSD Treatment in Persons Suffering From Anxiety Symptoms in Severe Somatic Diseases or in Psychiatric Anxiety Disorders
Acronym: LSD-assist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC 2016-00992
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Patients; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind, placebo-controlled, crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo, LSD (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo or lysergic acid diethylamide (LSD)
  Interventions: Drug: Placebo
- LSD, Placebo (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo or lysergic acid diethylamide (LSD)
  Interventions: Drug: LSD

INTERVENTIONS:
Drug: LSD — Lysergic Acid Diethylamide
  200ug per os, single dose
  Arms: LSD, Placebo
Drug: Placebo — Capsules containing mannitol looking identical to LSD
  Arms: Placebo, LSD

SUMMARY:
Background: Lysergic acid diethylamide (LSD) was extensively investigated in humans in the 1950s and 1960s. Particularly, LSD attenuated anxiety in patients with cancer. Clinical research with LSD ended in the 1970s due to regulatory restrictions but its use for personal and recreational purposes continued. In recent years, there has been a renewed interest in the use hallucinogens in psychiatric research and practices. LSD and psilocybin were reused in experimental studies in healthy subjects and in the treatment for anxiety in patients with life-threatening diseases. Specifically, a pilot study documented that LSD can be used safely and may reduce anxiety in these patients. Larger well-designed and placebo-controlled studies are warranted. Similar studies have recently been completed with the hallucinogen psilocybin.

Objective: To test the efficacy of LSD in patients with anxiety with or without life-threatening diseases.

Design: Double-blind, placebo-controlled random-order cross-over trial using two LSD (200 µg) and two placebo sessions with subjects acting as their own control.

Participants: 40 patients aged > 25 years with anxiety disorder (according to DSM-IV or a state-trait anxiety inventory score >40 in the STAI trait or state scale) with or without life-threatening illness.

Main outcome measures: Reduction in anxiety (STAI), depression (Hamilton depression rating scale, HDRS and Beck depression inventory, BDI), and general psychopathological symptoms (Symptom Check List 90 items, SCL-90) at 2, 8, and 16 weeks after LSD- compared with placebo-assisted psychotherapy.

Significance: Anxiety disorder (alone or in the context of life-threatening illness) is frequent and often insufficiently managed with available medications. This study will evaluate the potential benefits of single treatments with LSD in anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 25 years.
2. Meet DSM-IV criteria for anxiety disorder as indicated by the Structured Clinical Interview for the DSM (SCID)-IV or have a score of at least 40 on the state- or trait STAI scale at study inclusion.
3. 40% or more of the participants should have a diagnosis of advanced-stage potentially fatal illness (autoimmune, neurological, or cancer without central nervous system (CNS) involvement). Patients should be ambulatory and not terminal and likely to have a roughly estimated life expectancy of > twelve months.
4. Patients without advanced-stage potentially fatal illness need to meet DSM-IV criteria for anxiety disorder (elevated STAI score not sufficient for inclusion)
5. Sufficient understanding of the study procedures and risks associated with the study.
6. Participants must be willing to adhere to the study procedures and sign the consent form.
7. Participants are willing to refrain from taking any psychiatric medications during the experimental session period. If they are being treated with antidepressants or are taking anxiolytic medications on a fixed daily regimen such drugs must be discontinued long enough before the LSD/placebo treatment session to avoid the possibility of a drug-drug interaction (the interval will be at least 5 times the particular drug's half-life [typically 3-7 days]).
8. If in ongoing psychotherapy, those recruited into the study may continue to see their outside therapist, provided they sign a release for the investigators to communicate directly with their therapist. Participants should not change therapists, increase or decrease the frequency of therapy or commence any new type of therapy during the study (not including the follow-up).
9. Participants must also refrain from the use of any psychoactive drugs, with the exception of the long term pain medication or caffeine or nicotine, within 24 hours of each LSD/placebo treatment session. They must agree not to use nicotine for at least 2 hours before and 6 hours after each dose of LSD. They must agree to not ingest alcohol-containing beverages for at least 1 day before each LSD treatment session. Non-routine medications for treating breakthrough pain taken in the 24 hours before the LSD treatment session may result in rescheduling the treatment session to another date, with the decision at the discretion of the investigators after discussion with the participant.
10. Participants must be willing not to drive a traffic vehicle or to operate machines within 24 h after LSD/placebo administration.

Exclusion Criteria:

1. Women who are pregnant or nursing, or of child bearing potential and are not practicing an effective means of birth control (double-barrier method, i.e. pill/intrauterine device and preservative/diaphragm).
2. Past or present diagnosis of a primary psychotic disorder. Subjects with a first degree relative with psychotic disorders are also excluded.
3. Past or present bipolar disorder (DSM-IV)
4. Current substance use disorder (within the last 2 months, DSM-V, except nicotine)
5. Somatic disorders including central nervous system (CNS) involvement of the cancer, severe cardiovascular disease, untreated hypertension, severe liver disease (liver enzymes increase by more than 5 times the upper limit or normal) or severely impaired renal function (estimated creatinine clearance <30 ml/min), or other that in the judgement of the investigators pose too great potential for side effects
6. Weight < 45 kg
7. Suicide risk or likely to require psychiatric hospitalization during the course of the study
8. Requiring ongoing concomitant therapy with a psychotropic drug (other than as needed, anxiety medications, and pain control medications) and unable or unwilling to comply with the washout period.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Reduction in anxiety assessed by questionnaires | 16 weeks post-intervention
  Reduction in anxiety assessed by questionnaires (STAI) 16 weeks after LSD compared with placebo

SECONDARY OUTCOMES:
Reduction in Depression assessed by questionnaires | 2, 8 and 16 weeks post-intervention
  Reduction in depression will be assessed by questionnaires (HDRS, BDI) 2, 8 and 16 weeks after LSD compared with placebo
Reduction in anxiety assessed by questionnaires | 2 and 8 weeks post-intervention
  Reduction in anxiety will be assessed by questionnaire (STAI) 2 and 8 weeks after LSD compared with placebo
Reduction of psychopathological symptoms assessed by questionnaires | 2, 8 and 16 weeks post-intervention
  Reduction of psychopathological symptoms will be assessed by questionnaire (SCL-90) 2, 8, and 16 weeks after LSD compared with placebo
Sustained Response assessed by questionnaires | 52 weeks post intervention
  Follow-up using different questionnaires to compare (within-subject) the 52-week response with Responses from baseline and 16-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gasser, MD, Principal Investigator — Private Practice
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Private Practice P.Gasser, Solothurn, Canton of Solothurn

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holze F, Gasser P, Muller F, Dolder PC, Liechti ME. Lysergic Acid Diethylamide-Assisted Therapy in Patients With Anxiety With and Without a Life-Threatening Illness: A Randomized, Double-Blind, Placebo-Controlled Phase II Study. Biol Psychiatry. 2023 Feb 1;93(3):215-223. doi: 10.1016/j.biopsych.2022.08.025. Epub 2022 Sep 5. PMID 36266118